CLINICAL TRIAL: NCT06624254
Title: Ventilator Mode and Respiratory Physiology
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Alex Pearce, Principal Investigator, University of California, San Diego
Other Study IDs: 807319
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Pulmonary Disease; Respiratory Failure; Respiratory Effort; Breathing Mechanics
MeSH Terms: conditions — Lung Diseases; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adaptive Pressure Control: On adaptive pressure control mode with acute respiratory failure
  Interventions: Other: lung mechanics, respiratory drive and effort

INTERVENTIONS:
Other: lung mechanics, respiratory drive and effort — Patient lung mechanics and respiratory drive and effort will be measured

SUMMARY:
Modern intensive care units (ICUs) are increasingly adopting newer modes of mechanical ventilation such as adaptive pressure control (APC) modes but there are limited data available regarding risks and benefits of newer modes versus traditional ventilation modes. APC can inadvertently deliver high tidal volumes, which maybe harmful. High tidal volumes may be unrecognized by the provider, due to the complexities of ventilator algorithms and patient interactions. The objective of this aim is to identify risk factors for excess tidal volumes in patients on adaptive pressure control.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to ICU with acute respiratory failure
* On adaptive pressure control mode of ventilation
* Tidal volumes set between 5-8 cc/kg ideal body weight

Exclusion Criteria:

* Current use of neuromuscular blockade
* Inability to obtain consent from patient or surrogate decision maker
* Treating clinician refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Human subjects admitted to the intensive care unit requiring invasive mechanical ventilation for acute respiratory failure on adaptive pressure control modes of ventilation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-21 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Excess tidal volume | From enrollment to end of monitoring at 4 hours
  Exhaled tidal volume greater than 2cc/kg ideal body weight above intended or set tidal volume

CONTACTS AND LOCATIONS:
Overall Officials: Alex Pearce, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego Health, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
reasonable requests for IPD will be considered by the investigators